CLINICAL TRIAL: NCT04756648
Title: An Open, Dose Escalation/Dose Exploration, Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single/Multiple Infusion of CT0180 Injection in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Phase I Clinical Trial of CT0180 Cells in the Treatment of Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT0180-CG1203
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Advanced Hepatocellular Carcinoma; CT0180 Cells; GPC3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CT0180 cells (Experimental): CT0180 Cells infusion after lymphocyte-depleting with fludarabine and cyclophosphamide.
  Interventions: Drug: CT0180 Cells

INTERVENTIONS:
Drug: CT0180 Cells — Five dose levels were tentatively determined.
  Other Names: CT0180 humanized anti GPC3 autogenous T Cell injection

SUMMARY:
A Phase I Clinical Study ofCT0180 cells in Patients with Advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
Primary objectives:

Evaluate the safety and tolerance of CT0180 cells in patients with advanced hepatocellular carcinoma within 28 days after the first infusion

Secondary objectives:

* Evaluate the metabolic kinetics of CT0180 cells ; · Evaluate overall safety and tolerability ; · Evaluate the initial efficacy of CT0180 cell infusion in the treatment of advanced hepatocellular carcinoma with positive Glypican-3（GPC3 ）expression.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years, either sex；
2. Patients with clinically or pathologically confirmed hepatocellular carcinoma were treated with surgery or local treatment It is not suitable for surgery or local radical treatment;
3. Progression or intolerance after at least one previous systemic treatment, or due to specific reasons unable to receive systemic treatment. Systemic therapy can include: Programmed Death 1（PD-1） / programmed cell death-Ligand 1（PD-L1） monoclonal antibody Antibodies, molecular targeted drugs (e.g. sorafenib, regofinib, renvastinib)and conventional chemotherapy, etc;
4. According to Barcelona Clinic Liver Cancer（BCLC）, the patients are classified into Grade C or Grade B unsuitable for local treatment/progressive disease after local treatment;
5. In tumor tissue samples GPC3 is detected positive by immunohistochemistry (IHC);
6. According to Response Evaluation Criteria in SolidTumors（RECIST1.1）,patients have at least one evaluable target lesion, defined as: the longest diameter of non-lymph node lesion ≥ 10 mm, or the shortest diameter of lymph node lesion ≥ 15 mm); hepatic lesions require arterial phase contrast enhancement;
7. Expected survival is > 12 weeks;
8. Cirrhosis status Child-Pugh score: Grade A;
9. Eastern Cooperative Oncology Group（ ECOG） Performance Status score: 0 to 1 point;
10. If the patient is HBsAg positive or HBcAb positive, HBV-DNA should be <2000 IU/ml. HBsAg positive patients must receive antiviral treatment ;
11. Acceptable routine blood test showing no contraindication to the lymphodepletion pretreatment and adequate liver, renal, cardiovascular, respiratory function;
12. Have venous accesses for apheresis;
13. Subjects of childbearing age must undergo a serum pregnancy test within 14 days before the initiation of the study and the result must be negative. In addition, they should be willing to use a reliable method of contraception during the trial (within 52 weeks after cell infusion); male subjects whose spouses are women of childbearing age should undergo sterilization surgery or agree to use a reliable method of contraception during the trial;
14. Understand and sign informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. Hepatitis virus C antibodies ,human immunodeficiency virus（HIV） antibodies or Syphilis Serological tests are positive;
3. Any uncontrol active infection, including but not limited to active tuberculosis;
4. Have clinically significant thyroid dysfunction except the stable control after treatment;
5. Previous or present hepatic encephalopathy;
6. Current clinically significant ascites;
7. Imaging results:≥50% of the liver is replaced by tumor or portal vein main tumor thrombus, or metastases to the central nervous system, or tumor thrombus invasion of mesenteric vein / inferior vena cava;
8. Patients with a history of organ transplantation or waiting for organ transplantation (including liver transplantation);
9. The side effects caused by the previous treatment of the subjects did not return to Common Terminology Criteria for Adverse Events（CTCAE） ≤1; except hair loss and other tolerable events determined by investigator;
10. Patients who had received systemic steroids or other immunosuppressive agents within 7 days before apheresis, except inhaled steroids;
11. History of severe allergy ,allergic to CT0180 cell fluid adjuvant such as Dimethyl sulfoxide（DMSO）;
12. Has signs of central nervous system disease or an abnormal neurological examination with clinical significance;
13. Subjects with unstable or active ulcers, gastrointestinal bleeding, or pump inhibitor intolerance;
14. Patients with a history of organ transplantation or waiting for organ transplantation;
15. Previously received anti-PD-1/ PD-L1 monoclonal antibody therapy within 4 weeks or local treatment and systemic chemotheray within 2 weeks or immunotheray and molecular targeted drugs within 1 week before apheresis;
16. Previously received GPC3 targeted therapy;
17. Major surgery or significant trauma occurred within 4 weeks before apheresis, or it is expected that major surgery needs to be performed during the trial;
18. Patients who had incurable malignant tumors in the past 5 years or at the same time, except cervical cancer in situ and basal cell carcinoma of skin;
19. Other serious diseases that may restrict the subjects from participating in the trial ；
20. The researcher assessed that the subjects were unable or unwilling to comply with the requirements of the trial protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity（DLT） | 28 days
  Safety
Maximal Tolerable Dose（MTD） | 28 days
  tolerability evaluation
Adverse Event（AE） | 28 days
  Incidence rate
Adverse Event of Special Interest （ AESI） | 28 days
  Incidence rate

SECONDARY OUTCOMES:
Number of cells | 52 weeks
  Pharmacokinetics is the "Implantation endpoint" which is defined as the number of copies of the CT0180 DeoxyriboNucleic Acid（DNA）in peripheral blood detected at each visit after infusion until any two consecutive test results are negative or below the detection limit. Duration of CT0180 Cell persistence is the period from the day of infusion to the first negative test result or result lower than the detection limit
Treatment Emergent Adverse Event(TEAE) | 52 weeks
  Incidence rate
Antitumor efficacy-Objective response rate (ORR) | 52 weeks
  The number of cases in which tumor size is reduced to partial response (PR) or complete response (CR) / the total number of evaluable cases (%). In the event of partial response( PR) or complete response (CR), the subjects should confirm it no less than 4 weeks after the first evaluation
Antitumor efficacy-Duration of response (DOR) | 52 weeks
  The period from the first evaluation of complete response ( CR) or partial response (PR) to the first evaluation of progressive disease (PD)or death of any cause.
Antitumor efficacy-Progression-free survival (PFS) | 52 weeks
  The period from the day when the subject receives the first study treatment to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first
Antitumor efficacy-Overall survival (OS) | 52 weeks
  The period from the first study treatment to any cause of death
Antitumor efficacy-Disease control rate (DCR) | 52 weeks
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).
Antitumor efficacy-Duration of disease control (DDC) | 52 weeks
  The period from the first evaluation of CR, PR, or SD to the first evaluation of PD or any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No